CLINICAL TRIAL: NCT02120417
Title: A Randomized, Double-Blind, Phase 2 Study of Ruxolitinib or Placebo in Combination With Capecitabine in Subjects With Advanced or Metastatic HER2-Negative Breast Cancer
Brief Title: A Study of Ruxolitinib in Combination With Capecitabine in Subjects With Advanced or Metastatic HER2-negative Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated as other related studies of ruxolitinib did not provide sufficient efficacy to warrant continuation.
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INCB 18424-268
Record Dates: First submitted 2014-04-18; First posted 2014-04-22 (Estimated); Results first posted 2017-07-12 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-01

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — ruxolitinib; Capecitabine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment A - Capecitabine and ruxolitinib (Experimental)
  Interventions: Drug: Ruxolitinib; Drug: Capecitabine
- Treatment B - Capecitabine and placebo (Active Comparator)
  Interventions: Drug: Capecitabine; Drug: Placebo

INTERVENTIONS:
Drug: Ruxolitinib — 5 mg tablets to be administered by mouth
  Ruxolitinib 15 mg BID (starting dose)
  Other Names: Jakafi ®; Jakavi ®
  Arms: Treatment A - Capecitabine and ruxolitinib
Drug: Capecitabine — Capecitabine 2000 mg/m^2 daily given as 1000 mg/m^2 twice a day (BID) (starting dose) Day 1-14 of each 21 day cycle
Drug: Placebo — 5 mg matching placebo tablets to be administered by mouth
  Arms: Treatment B - Capecitabine and placebo

SUMMARY:
This was a randomized, double-blind, placebo-controlled phase 2 clinical trial comparing the overall survival of women with advanced or metastatic HER2-negative breast cancer who received treatment with capecitabine in combination with ruxolitinib versus those who received treatment with capecitabine alone.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed HER2-negative adenocarcinoma of the breast
* Locally advanced (Stage 3B) or metastatic (Stage 4) disease
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2
* Received up to 2 prior chemotherapy regimens (not including neoadjuvant/adjuvant therapy) for advanced or metastatic disease
* Participants with hormone-receptor positive tumors must have failed available lines of hormonal therapy unless hormone therapy was not tolerated or not clinically appropriate
* ≥ 2 weeks elapsed from the completion of previous treatment regimen and must have recovered or be at a new stable baseline from any related toxicities
* Radiographically measurable or evaluable disease
* An mGPS of 1 or 2 as defined below:

  * Criteria:

    1. modified Glasgow prognostic score (mGPS) of 1: CRP > 10 mg/L and albumin ≥ 35 g/L
    2. mGPS of 2: C-reactive protein (CRP) > 10 mg/L and albumin < 35 g/L

Exclusion Criteria:

* Received prior treatment with capecitabine or fluoropyrimidine for advanced or metastatic disease
* Received more than 2 prior regimens for advanced or metastatic disease (not including hormonal therapy in the metastatic setting or neoadjuvant or adjuvant therapies)
* Unknown hormone-receptor status
* Ongoing radiation therapy or radiation therapy administered within 2 weeks of enrollment
* Concurrent anticancer therapy
* Inadequate renal, hepatic or bone marrow function
* Another current or previous malignancy within 2 years of study entry unless approved by the sponsor

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Kennealey, MD, Study Director — Incyte Corporation
Locations (106):
- United States (80):
  - Birmingham, Alabama
  - Chandler, Arizona
  - Sedona, Arizona
  - La Jolla, California
  - Los Angeles, California
  - Oxnard, California
  - San Diego, California
  - San Francisco, California
  - Santa Monica, California
  - Aurora, Colorado
  - Denver, Colorado
  - New Haven, Connecticut
  - Washington D.C., District of Columbia
  - Fort Myers, Florida
  - Hialeah, Florida
  - Miami, Florida
  - Plantation, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Marietta, Georgia
  - Savannah, Georgia
  - Chicago, Illinois
  - Quincy, Illinois
  - Springfield, Illinois
  - Urbana, Illinois
  - Ames, Iowa
  - Wichita, Kansas
  - Louisville, Kentucky
  - Baton Rouge, Louisiana
  - Baltimore, Maryland
  - Detroit, Michigan
  - Kalamazoo, Michigan
  - Duluth, Minnesota
  - Minneapolis, Minnesota
  - Kansas City, Missouri
  - St Louis, Missouri
  - Grand Island, Nebraska
  - Omaha, Nebraska
  - Camden, New Jersey
  - Hackensack, New Jersey
  - Farmington, New Mexico
  - Albany, New York
  - Johnson City, New York
  - New York, New York
  - The Bronx, New York
  - Goldsboro, North Carolina
  - Pinehurst, North Carolina
  - Canton, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Middletown, Ohio
  - Portland, Oregon
  - Bethlehem, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Greenville, South Carolina
  - Chattanooga, Tennessee
  - Germantown, Tennessee
  - Nashville, Tennessee
  - Arlington, Texas
  - Bedford, Texas
  - Dallas, Texas
  - El Paso, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - McAllen, Texas
  - Plano, Texas
  - Tyler, Texas
  - Ogden, Utah
  - Salt Lake City, Utah
  - Fairfax, Virginia
  - Norfolk, Virginia
  - Richmond, Virginia
  - Salem, Virginia
  - Seattle, Washington
  - Green Bay, Wisconsin
  - Milwaukee, Wisconsin
- France (2):
  - La Roche-sur-Yon
  - Paris
- Italy (9):
  - Alba
  - Fano
  - Foggia
  - Lecco
  - Milan
  - Naples
  - Pontedera
  - Roma
  - Saronno
- Lisbon, Portugal
- Spain (5):
  - A Coruña
  - Barcelona
  - Jaén
  - Lleida
  - Madrid
- United Kingdom (9):
  - Cardiff
  - Glasgow
  - Kingston upon Thames
  - London
  - Nottingham
  - Sutton
  - Taunton
  - Truro
  - Yeovil

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 72 study centers (65 in the United States and 7 in the European Union [3 in the United Kingdom, 3 in Spain, and 1 in Portugal]).
Groups:
- Treatment A - Capecitabine and Ruxolitinib: Capecitabine given as 1000 mg/m^2 twice a day (BID) on day 1 to day 14 of each 21-day cycle with the addition of Ruxolitinib 15 mg (three 5 mg tablets) BID to be administered by mouth on day 1 to day 21 of each 21-day cycle
- Treatment B - Capecitabine and Placebo: Capecitabine given as 1000 mg/m^2 twice a day (BID) on day 1 to day 14 of each 21-day cycle with the addition of 15 mg (three 5 mg tablets) matching placebo BID to be administered by mouth on day 1 to day 21 of each 21-day cycle
Period: Overall Study
Arm/Group | Treatment A - Capecitabine and Ruxolitinib | Treatment B - Capecitabine and Placebo
Started (Overall Number of Participants Analyzed) | 76 | 73
Completed (Number of participants remaining on treatment at the 08 FEB 2016 data cutoff.) | 16 | 5
Not Completed | 60 | 68
Not completed — Death | 5 | 1
Not completed — Adverse Event | 3 | 9
Not completed — Participant decision | 4 | 4
Not completed — Disease progression | 41 | 45
Not completed — Noncompliance with study treatment | 0 | 2
Not completed — Physician Decision | 2 | 3
Not completed — Other unspecified | 5 | 4

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) population consisted of all participants randomized to the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment A - Capecitabine and Ruxolitinib | Treatment B - Capecitabine and Placebo | Total
Number analyzed (Participants) | 76 | 73 | 149
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (11.00) | 55.0 (12.75) | 54.6 (11.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 73 | 149
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall survival is reported here by the number of days from randomization to death until the data cutoff for the final analysis. The hazard ratio (80% CI) for ruxolitinib versus placebo was estimated using a Cox regression model stratified by hormone-receptor status.
Time Frame: Randomization until death due to any cause up to 19 months or the data cutoff 08FEB2016.
Population: The Intent-to-Treat (ITT) population consisted of all participants randomized to the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A - Capecitabine and Ruxolitinib | Treatment B - Capecitabine and Placebo
Number analyzed (Participants) | 76 | 73
Participants
  Death events | 39 | 38
  Censored events | 37 | 35
Statistical Analysis 1: Comparison: Treatment A - Capecitabine and Ruxolitinib vs Treatment B - Capecitabine and Placebo; Test type: Superiority or Other; p = 0.762, Log Rank; The P-value was analyzed by Log-Rank Test stratified by Hormone Receptor Status; Hazard Ratio (HR) = 0.932, 80% CI 2-sided [0.694 to 1.252]

2. Primary Outcome: Median Survival
Description: Survival was assessed by the time to death or censoring up until 08Feb2016. Participants with no observed death were treated as right-censored at their last date known to be alive. The survival time was analyzed using the Kaplan-Meier method.
Time Frame: Randomization until death due to any cause up to 19 months or the data cutoff 08FEB2016.
Population: The Intent-to-Treat (ITT) population consisted of all participants randomized to the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment A - Capecitabine and Ruxolitinib | Treatment B - Capecitabine and Placebo
Number analyzed (Participants) | 76 | 73
months | 11.2 [7.5 to 12.7] | 10.9 [6.0 to 13.1]

3. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival was defined as the time from the randomization date to the earliest date of disease progression, as measured by investigator assessment of objective radiographic disease assessments per RECIST (v1.1), or death from any cause if earlier. Progression-free survival time distribution and median survival for each treatment group were analyzed using the Kaplan-Meier method.
Time Frame: Randomization to disease progression, or death due to any cause if sooner up to 19 months or the data cutoff 08FEB2016.
Population: The Intent-to-Treat (ITT) population consisted of all participants randomized to the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment A - Capecitabine and Ruxolitinib | Treatment B - Capecitabine and Placebo
Number analyzed (Participants) | 76 | 73
months | 4.5 [2.3 to 6.1] | 2.5 [2.1 to 4.1]

4. Secondary Outcome: Percentage of Participants Achieving Objective Response Rate
Description: Objective response rate determined by radiographic disease assessments per RECIST (v1.1), by investigator assessment and was defined as the percentage of participants with Complete Response (CR) or Partial Response (PR) by Response Evaluation Criteria in Solid Tumours (RECIST) at any post baseline visit. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST) for target lesions and assessed by computed tomography (CT) and/or magnetic resonance imaging (MRI) : Complete Response (CR), Disappearance of all target and non-target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions with no worsening of non-target lesions and no new lesions; Overall Response (OR) = CR + PR.
Time Frame: Randomization through end of study up to 19 months or the data cutoff 08FEB2016.
Population: The Intent-to-Treat (ITT) population consisted of all participants randomized to the study.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment A - Capecitabine and Ruxolitinib | Treatment B - Capecitabine and Placebo
Number analyzed (Participants) | 76 | 73
percentage of participants
  Complete Response rate | 0.0 | 0.0
  Partial Response rate | 28.9 | 13.7

5. Secondary Outcome: Duration of Response (DOR)
Description: The DOR was defined as the difference (in number of months) between the end of response and the start of response for participants who had at least 1 response measurement. The start of a response was the first visit where the participant achieved a partial response or better based on RECIST (v1.1) criteria. The end of response was the earlier of death or progressive disease based on RECIST (v1.1) criteria. The date of progressive disease was the date on which progression was first recorded. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST) for target lesions and assessed by computed tomography (CT) and/or magnetic resonance imaging (MRI) : Complete Response (CR), Disappearance of all target and non-target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions with no worsening of non-target lesions and no new lesions; Overall Response (OR) = CR + PR.
Time Frame: Randomization through end of study up to 19 months or the data cutoff 08FEB2016.
Population: The Intent-to-Treat (ITT) population consisted of all participants randomized to the study.
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Treatment A - Capecitabine and Ruxolitinib | Treatment B - Capecitabine and Placebo
Number analyzed (Participants) | 76 | 73
months | 4.2 [3.5 to 4.6] | 4.4 [3.8 to 6.4]

6. Secondary Outcome: Percentage of Participants Achieving Clinical Benefit Rate
Description: Clinical benefit rate was defined as a complete response, partial response, or stable disease, determined by investigator assessment of objective radiographic disease assessments per RECIST (v1.1) that lasted for ≥ 6 months. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST) for target lesions and assessed by computed tomography (CT) and/or magnetic resonance imaging (MRI) : Complete Response (CR), Disappearance of all target and non-target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions with no worsening of non-target lesions and no new lesions; Overall Response (OR) = CR + PR.
Time Frame: Randomization through end of study up to 19 months or the data cutoff 08FEB2016.
Population: The Intent-to-Treat (ITT) population consisted of all participants randomized to the study.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment A - Capecitabine and Ruxolitinib | Treatment B - Capecitabine and Placebo
Number analyzed (Participants) | 76 | 73
percentage of participants | 13.2 | 6.8

7. Primary Outcome: Percentage of Participants Achieving Overall Survival
Description: Overall survival was assessed by the time to death or censoring up until 08Feb2016. Participants with no observed death were treated as right-censored at their last date known to be alive. The survival time was analyzed using the Kaplan-Meier method.
Time Frame: Randomization until death due to any cause at month 3, 6, 9, 12 and 15 or the data cutoff 08FEB2016.
Population: The Intent-to-Treat (ITT) population consisted of all participants randomized to the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment A - Capecitabine and Ruxolitinib | Treatment B - Capecitabine and Placebo
Number analyzed (Participants) | 76 | 73
percentage of participants
  Month 3 Survival Rate | 0.855 [0.753 to 0.917] | 0.750 [0.633 to 0.835]
  Month 6 Survival Rate | 0.674 [0.554 to 0.769] | 0.635 [0.511 to 0.735]
  Month 9 Survival Rate | 0.537 [0.404 to 0.652] | 0.546 [0.417 to 0.657]
  Month 12 Survival Rate | 0.435 [0.289 to 0.573] | 0.427 [0.286 to 0.561]
  Month 15 Survival Rate | 0.319 [0.174 to 0.475] | 0.294 [0.148 to 0.456]

ADVERSE EVENTS:
Time Frame: Participants received study treatment in continuous 21-day cycles until they met withdrawal criteria up to 19 months or the data cutoff 08FEB2016. The cutoff date of 08Feb2016 was chosen based on the date that the sponsor became aware that the seventieth death had occurred in the randomized population.
Description: The safety evaluable population consisted of all participants enrolled in the study who received at least 1 dose of any study treatment (ie, ruxolitinib, placebo, or capecitabine).
  Adverse events were collected from participants and tabulated by the MedDRA version 17.0 preferred term and system organ class (SOC).The intensity and whether treatment related was tabulated and reported by the investigator.
Arm/Group | Treatment A - Capecitabine and Ruxolitinib | Treatment B - Capecitabine and Placebo
Serious Adverse Events (participants affected / at risk) | 28/71 | 29/71
Other Adverse Events (participants affected / at risk) | 69/71 | 69/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A - Capecitabine and Ruxolitinib (N=71) | Treatment B - Capecitabine and Placebo (N=71)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 2
Colitis (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 5 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 4
Non-cardiac chest pain (General disorders) | 2 | 1
Oedema (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 2
Hepatic failure (Hepatobiliary disorders) | 2 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Clostridium difficile infection (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 1
Sepsis (Infections and infestations) | 2 | 2
Urinary tract infection (Infections and infestations) | 2 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 3 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Metabolic disorder (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Embolic stroke (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 2
Syncope (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 6
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Deep vein thrombosis (Vascular disorders) | 0 | 3
Embolism (Vascular disorders) | 1 | 2
Hypertension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A - Capecitabine and Ruxolitinib (N=71) | Treatment B - Capecitabine and Placebo (N=71)
Anaemia (Blood and lymphatic system disorders) | 35 | 18
Neutropenia (Blood and lymphatic system disorders) | 9 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 1
Tachycardia (Cardiac disorders) | 6 | 3
Abdominal distension (Gastrointestinal disorders) | 5 | 6
Abdominal pain (Gastrointestinal disorders) | 12 | 6
Constipation (Gastrointestinal disorders) | 18 | 17
Diarrhoea (Gastrointestinal disorders) | 33 | 19
Dyspepsia (Gastrointestinal disorders) | 6 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 4
Nausea (Gastrointestinal disorders) | 39 | 35
Stomatitis (Gastrointestinal disorders) | 19 | 12
Vomiting (Gastrointestinal disorders) | 26 | 19
Fatigue (General disorders) | 40 | 31
Oedema (General disorders) | 4 | 3
Pyrexia (General disorders) | 12 | 10
Oedema peripheral (General disorders) | 10 | 14
Upper respiratory tract infection (Infections and infestations) | 4 | 2
Urinary tract infection (Infections and infestations) | 6 | 6
Alanine aminotransferase increased (Investigations) | 6 | 4
Aspartate aminotransferase increased (Investigations) | 9 | 5
Blood alkaline phosphatase increased (Investigations) | 5 | 4
Blood creatinine increased (Investigations) | 5 | 3
Lymphocyte count decreased (Investigations) | 4 | 2
Neutrophil count decreased (Investigations) | 6 | 2
Platelet count decreased (Investigations) | 6 | 0
Weight decreased (Investigations) | 4 | 5
Weight increased (Investigations) | 6 | 4
White blood cell count decreased (Investigations) | 7 | 1
Decreased appetite (Metabolism and nutrition disorders) | 21 | 19
Dehydration (Metabolism and nutrition disorders) | 11 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 8 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 10 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 5
Dizziness (Nervous system disorders) | 13 | 13
Dysgeusia (Nervous system disorders) | 1 | 5
Headache (Nervous system disorders) | 16 | 9
Hypoaesthesia (Nervous system disorders) | 4 | 4
Neuropathy peripheral (Nervous system disorders) | 3 | 5
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 5
Anxiety (Psychiatric disorders) | 1 | 6
Insomnia (Psychiatric disorders) | 8 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 22 | 20
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 5
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 33 | 27
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 6 | 2
Hot flush (Vascular disorders) | 4 | 1
Hypertension (Vascular disorders) | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.